CLINICAL TRIAL: NCT03604887
Title: Umbilical Cord Length Index as a New Ultrasonographic Method for Prediction of Cord Abnormalities Before Delivery
Brief Title: Umbilical Cord Length Index for Prediction of Cord Abnormalities Before Delivery
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: UCLI
Record Dates: First submitted 2018-07-21; First posted 2018-07-30 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Umbilical Cord Problem
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: All pregnant women who will attend the labor unit during the study period will be invited to participate in the study.
  Interventions: Diagnostic Test: ultrasonography

INTERVENTIONS:
Diagnostic Test: ultrasonography — Ultrasound evaluation will be done with transducer abdominal probe. The amount of amniotic fluid and umbilical cord sections will be determined by evaluating the images obtained from the sagittal plane in the ultrasound evaluations in the 4 abdominal quadrants.
  When the anatomical structure of the umbilical cord is considered, it is folded in amniotic fluid. The folds appear as umbilical cord rings, side-by-side at the sagittal sections.
  Scoring of "umbilical cord length index"
  * 1 point will be given for each quadrant where the umbilical cord was observed.
  * 0.5 point will be given for each umbilical cord ring in one quadrant. Every quadrant will be evaluated in this manner, and the total score will be calculated.

SUMMARY:
The umbilical cord plays an essential role in intrauterine life. It is the pathway between mother, placenta and fetus during pregnancy and delivery. Complete cord occlusion often leads to fetal demise, while intermittent occlusion has been associated with intrauterine brain damage. Compression and vasospasm in utero are important factors in fetal distress. Nuchal Umbilical Cord can be diagnosed antepartum using ultrasound, but the complications are unpredictable and unpreventable

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* Pregnant ≥ 37 weeks gestation.
* Women who will accept to participate in the study

Exclusion Criteria:

* Preterm deliveries.
* Amniotic fluid abnormalities (oligohydramnios, polyhydramnios).
* Intrauterine growth retardation
* Early membrane rupture
* Women need urgent cesarean section.
* Multifetal gestation.
* Placenta previa.
* Fetuses with major congenital anomalies.
* Women with chronic maternal illness as hypertension

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are in labor will be followed up through regular fetal heart rate monitoring and clinically using partograph to monitor the progress of labor. Fetal heart rate changes and cases with abnormal progress of labor will be recorded. Mode of delivery either vaginal or cesarean will be noted. Those who are scheduled for elective CS will be evaluated during and after cesarean section.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
The sensitivity of "Umbilical cord length index" in diagnosis of long and short umbilical cords. | 15 minutes
  Ultrasonographic scoring of umbilical cord length

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No